CLINICAL TRIAL: NCT04095104
Title: Adjunctive Anti-Obesity Pharmacotherapy in Adolescents and Young Adults After Bariatric Surgery: A Randomized Controlled Pilot Study
Brief Title: Adjunct Phentermine + Topiramate After Bariatric Surgery in 12-24 Year Olds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Colorado- Clinical and Translational Sciences Institute (Unknown); University of Colorado- Nutrition Obesity Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-2793; 5P30DK048520-24 (NIH)
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Obesity, Morbid; Bariatric Surgery; Adolescent; Young Adult; Drug Therapy
Keywords: Pilot; Feasibility; Initial Efficacy; Randomized Controlled Trial
MeSH Terms: conditions — Obesity, Morbid | interventions — Phentermine; Topiramate

STUDY DESIGN:
Intervention Model Description: Two-arm parallel assignment where the experimental arm will receive active drugs + standard of care and the control arm will receive placebo drugs + standard of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: At baseline, each participant will be randomized 1:1 to either 12 weeks of phentermine, topiramate and standard of care or 12 weeks of phentermine placebo, topiramate placebo, and standard of care. This randomization will be blinded to the participant, investigator, care providers, and outcomes assessor for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phentermine & Topiramate (Experimental): Phentermine- Formulation: 8mg scored tablet, Dosage/Frequency/Duration:
  4mg x 7d then 8mg x 7d then 12mg x 7d then 16mg x 63d, taken once every morning
  +
  Immediate release topiramate- Formulation: 25mg tablet, Dosage/Frequency/Duration: 25mg x 7d then 50mg x 7d then 75mg x 7d then 100mg x 63d then 50mg x 7 days then 25mg x 7d, taken once every morning
  +
  Standard of Care (multidisciplinary postoperative bariatric surgery clinic visits)
  Interventions: Drug: Phentermine; Drug: Immediate Release Topiramate
- Placebo Drugs (Placebo Comparator): Placebo Phentermine- Formulation: 8mg scored tablet, Dosage/Frequency/Duration: 4mg x 7d then 8mg x 7d then 12mg x 7d then 16mg x 63d, taken once every morning
  +
  Placebo Immediate release topiramate- Formulation: 25mg tablet, Dosage/Frequency/Duration: 25mg x 7d then 50mg x 7d then 75mg x 7d then 100mg x 63d then 50mg x 7 days then 25mg x 7d, taken once every morning
  +
  Standard of Care (multidisciplinary postoperative bariatric surgery clinic visits)
  Interventions: Drug: Placebo for Phentermine; Drug: Placebo for Immediate Release Topiramate

INTERVENTIONS:
Drug: Phentermine — Phentermine tablet
  Other Names: Lomaira; Adipex-P; C045TQL4WP; 2-methyl-1-phenylpropan-2-amine
  Arms: Phentermine & Topiramate
Drug: Immediate Release Topiramate — Topiramate tablet
  Other Names: Topamax; 0H73WJJ391; [(3aS,5aR,8aR,8bS)-2,2,7,7-tetramethyl-5,5a,8a,8b-tetrahydrodi[1,3]dioxolo[4,5-a:5',3'-d]pyran-3a-yl]methyl sulfamate
  Arms: Phentermine & Topiramate
Drug: Placebo for Phentermine — Compounded tablet to mimic phentermine 8mg tablet
  Arms: Placebo Drugs
Drug: Placebo for Immediate Release Topiramate — Compounded tablet to mimic immediate release topiramate 25mg tablet
  Arms: Placebo Drugs

SUMMARY:
The goal of this pilot study is to establish the feasibility and initial efficacy of the combination of phentermine and topiramate for adolescents and young adults who require additional risk reduction after bariatric surgery. This study will use a randomized, placebo-controlled, double-blinded design to evaluate an adjunctive 12-week intervention of phentermine + topiramate + standard of care vs. placebos + standard of care 6 months after bariatric surgery, among 12 to 24 year olds who don't achieve expected weight loss or who remain severely obese (n=10 total).

ELIGIBILITY:
Inclusion Criteria:

* Status post sleeve gastrectomy or roux-en-y gastric bypass
* At 6 months after bariatric surgery, has not achieved >= 26% decrease in weight from preoperative weight (within 1 week of surgery) OR remains severely obese (>=120% of 95th%ile or BMI >=35kg/m2 for 12-17yo; BMI >=35kg/m2 for 18-24yo)

Exclusion Criteria:

* Absolute contraindication to phentermine or topiramate (i.e. phentermine:

history of coronary artery disease, stroke, arrhythmia, congestive heart failure, uncontrolled hypertension), hypersensitivity to sympathomimetic amines, current or recent (within 14 days) use of monoamine oxidase inhibitors, glaucoma, or hyperthyroidism; topiramate: hypersensitivity to topiramate, history of nephrolithiasis)

* Concomitant use of phenytoin, carbamazepine, or carbonic anhydrase inhibitors (e.g. zonisamide, acetazolamide, or dichlorphenamide)
* Use of anti-obesity medication within 6 months of screening
* Initiation of a new medication associated with weight loss or gain within 30 days of screening
* Type 2 diabetes mellitus
* Hypothalamic obesity
* Unmanaged (e.g. without medications and/or psychotherapy) clinically significant (determined by a mental health professional using diagnostic instruments and/or clinical interview) depression or anxiety
* History of any suicidal behavior within 30 days of screening or any suicidal ideation with either some intent to act or with intent and a specific plan within 30 days of screening
* History of schizophrenia
* Severe hepatic impairment (ALT >10x upper limit of normal or known synthetic liver dysfunction)
* Moderate or severe renal impairment (GFR <30mL/min/1.73m2)
* Dosage change to hypertension, dyslipidemia, depression, or anxiety medication <4 weeks prior to study enrollment
* Contraception started <7 days prior to study enrollment
* Current pregnancy/plans to become pregnant within 16 weeks from study drug start date
* Females without a long acting reversible contraceptive (LARC) who do not commit to using 2 forms of birth control

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime M Moore, MD, MPH, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in obesity. Data or samples shared will be coded, with no protected health information included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement. For more information or to submit a request, please contact clinicalresearchsupportcenter@ucdenver.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Phentermine & Topiramate: Participants were randomized to receive phentermine and topiramate plus standard post-bariatric care.
  Dosing schedule for active medication group:
  * Week 1: 4mg phentermine + 25mg immediate release topiramate
  * Week 2: 8mg phentermine + 50mg immediate release topiramate
  * Week 3: 12mg phentermine + 75mg immediate release topiramate
  Goal Dose:
  · Weeks 4-12: 16mg phentermine + 100mg immediate release topiramate
  Discontinuation (at study Visit 4):
  * Week 13: Discontinue Phentermine + Decrease topiramate to 50mg
  * Week 14: Decrease topiramate to 25mg for 7 days, then discontinue
  Notes:
  1. Participants who do not tolerate goal doses will be maintained at the highest tolerated dose.
  2. All topiramate and phentermine doses will be taken once daily in the morning.
- Placebo: Participants were randomized to receive placebo tablets that were compounded to look identical to phentermine and topiramate plus standard post-bariatric care.
  Dosing escalation, goal dose, and discontinuation for placebo group was identical to the active group.
Period: Overall Study
Arm/Group | Phentermine & Topiramate | Placebo
Started | 6 | 7
Completed | 6 | 6 (1 participant randomized to the placebo group withdrew before taking a single dose of study medication due to family psychosocial stressors unrelated to this study.)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phentermine & Topiramate: Participants were randomized to receive phentermine and topiramate plus standard post-bariatric care.
- Placebo: Participants were randomized to receive placebo tablets (compounded to look like phentermine and topiramate) plus standard post-bariatric care.
- Total: Total of all reporting groups
Arm/Group | Phentermine & Topiramate | Placebo | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Full Range); unit: years] | 16.7 [14 to 20] | 17.9 [15 to 20] | 17.3 [14 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 5 | 10
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: (Number enrolled divided by number eligible) x 100
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Groups:
- All Eligible Participants Before Randomization: The enrollment rate was calculated before randomization to active or placebo groups.
Arm/Group | All Eligible Participants Before Randomization
Number analyzed (Participants) | 68
percentage of participants | 19

2. Primary Outcome: Dropout Rate
Description: Number who do not complete the study divided by number enrolled
Time Frame: 24 months
Measure: Number; unit: percentage who withdrew among enrolled
Groups:
- Placebo: Participants were randomized to receive placebo tablets that were compounded to look like phentermine and topiramate plus standard post-bariatric care.
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 7
percentage who withdrew among enrolled | 0 | 7.7

3. Primary Outcome: Number of Participants Adherent to Study Drugs
Description: Presence of amphetamine in the urine at any study visit
Time Frame: 12 weeks
Population: The one participant randomized to the placebo group who withdrew before taking a single dose of study medication was not included in this outcome.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants were randomized to receive placebo tablets compounded to look like phentermine and topiramate plus standard post-bariatric care.
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
Participants | 5 | 0

4. Primary Outcome: Frequency of Adverse Events
Description: Unique adverse events documented prior to unblinding. Adverse events were elicited using a standardized checklist during study phone calls and in-person study visits, laboratory monitoring, review of systems, vitals, physical exam, and mood/suicidality assessment using validated instruments at every study visit.
Time Frame: 24 months
Population: as for outcome 3
Measure: Mean (Full Range); unit: unique adverse events per participant
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
unique adverse events per participant | 16 [10 to 27] | 8 [1 to 16]

5. Secondary Outcome: Percent BMI Change
Description: (Baseline BMI - BMI at 12 weeks)/Baseline BMI x 100
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: percent change
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
percent change | -3.61 [-13 to 2.86] | 1.89 [-0.06 to 4.62]

6. Secondary Outcome: Percent Weight Change
Description: (Baseline weight - weight at 12 weeks)/Baseline weight x 100
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: percent change
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
percent change | -4.72 [-12.14 to 2.61] | 0.83 [-6.94 to 6.47]

7. Secondary Outcome: Change in BMI Percent of the 95th%Ile
Description: (Baseline BMI % of the 95th%ile - BMI % of the 95th%ile at 12 weeks)
Time Frame: Baseline and 12 weeks
Population: For 1 member of the active group and 2 members of the placebo group, it was not appropriate to calculate a % above the 95th%ile either because BMI was <95th%ile or they were >19 completed years at the time point.
Measure: Mean (Full Range); unit: percentile change
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 5 | 4
percentile change | -6.2 [-19 to 4] | 2 [0 to 4]

8. Secondary Outcome: Change in Heart Rate
Description: (Heart rate at baseline - Heart rate at 12 weeks)
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: beats per minute
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
beats per minute | 2.89 [-16.67 to 47.33] | -0.83 [-16 to 6.33]

9. Secondary Outcome: Change in Systolic Blood Pressure
Description: Systolic blood pressure at baseline - Systolic blood pressure at 12 weeks
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
mmHg | 3.33 [-4 to 23] | 0.78 [-6.67 to 10]

10. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Diastolic blood pressure at baseline - Diastolic blood pressure at 12 weeks
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
mmHg | -1.33 [-20 to 11.67] | 4.17 [-6.67 to 20.67]

11. Secondary Outcome: Change in Total Cholesterol (mg/dL)
Description: Total cholesterol at baseline - Total cholesterol at 12 weeks
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
mg/dL | -18 [-47 to 33] | 6 [-16 to 37]

12. Secondary Outcome: Change in Triglycerides (mg/dL)
Description: Triglycerides at baseline - Triglycerides at 12 weeks
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
mg/dL | -7.17 [-42 to 55] | -6.33 [-71 to 47]

13. Secondary Outcome: Change in LDL Cholesterol (mg/dL)
Description: LDL at baseline - LDL at 12 weeks
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
mg/dL | -12.73 [-39 to 26.2] | 7.43 [0.2 to 21.6]

14. Secondary Outcome: Change in HDL Cholesterol (mg/dL)
Description: HDL at baseline - HDL at 12 weeks
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: mg/dL
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
mg/dL | -3.83 [-9 to 3] | -0.17 [-9 to 6]

15. Secondary Outcome: Change in Alanine Aminotransferase (ALT) (U/L)
Description: ALT at baseline - ALT at 12 weeks
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: U/L
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
U/L | 3.33 [-14 to 16] | 0.83 [-4 to 6]

16. Secondary Outcome: Change in Hemoglobin A1c (HbA1c) (%)
Description: HbA1c at baseline - HbA1c at 12 weeks
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: Percentage of glycated hemoglobin
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
Percentage of glycated hemoglobin | 0.05 [-0.3 to 0.7] | 0.10 [-0.1 to 0.3]

17. Secondary Outcome: Change in % Fat Mass
Description: % Fat mass at baseline - %Fat mass at 12 weeks measured by DEXA
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: percentage of fat mass
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
percentage of fat mass | -1.0 [-4.8 to 1.6] | 1.0 [-1.3 to 3.8]

18. Secondary Outcome: Change in Resting Metabolic Rate (RMR)
Description: RMR at baseline - RMR at 12 weeks measured by indirect calorimetry
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: kilocalories per day
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
kilocalories per day | -97.8 [-249.2 to 87] | -32.1 [-110.5 to 44.6]

19. Secondary Outcome: Change in Daily Kilocalorie Intake
Description: The average kilocalorie intake of 3 days was calculated each at baseline and 12 weeks. Kilocalories were calculated based on a standardized self-reported log of two weekdays and 1 weekend day.
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: kilocalories
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
kilocalories | -339.32 [-1409.39 to 412.08] | 94.85 [-266.99 to 719.63]

20. Secondary Outcome: Change in Hunger
Description: The adolescent/young adult will report subjective hunger before each meal and snack for 24 hours using a visual analogue slider scale (0= no hunger, 100 = most hunger) and this score will be averaged over the 24 hour period.
Time Frame: Baseline and 12 weeks
Population: VAS hunger ratings were missing from 1 participant in each the active and placebo groups
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | -10.76 [-36 to 11] | 0.20 [-39 to 44]

21. Secondary Outcome: Change in Satiety
Description: The adolescent/young adult will report subjective satiety 30 minutes after each meal and snack for 24 hours using a visual analogue slider scale (0= no fullness, 100 = most full) and this score will be averaged over the 24 hour period.
Time Frame: Baseline and 12 weeks
Population: VAS missing from 1 participant each in the active and placebo groups
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | -1.8 [-14 to 33] | -0.2 [-20 to 24]

22. Secondary Outcome: Change in Eating in the Absence of Hunger
Description: Validated questionnaire: Eating in the Absence of Hunger-Parent (EAH-P) completed by the parent/guardian about their adolescent/young adult. This measure has 14 items.
  Each item is on a 5-point Likert scale ranging from 1= "never" to 5= "always". A higher score indicates more eating in the absence of hunger.
  Total scores (minimum 14 to maximum 70) are calculated by taking the sum of the 14 items at each time point.
  The mean change in total scores by group are presented.
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | -7.3 [-23 to 0] | -0.5 [-5 to 7]

23. Secondary Outcome: Change in Cognitive Restraint
Description: The "Three-Factor Eating Questionnaire" will be completed by the adolescent/young adult. This is a 51-item questionnaire that assesses 3 eating behaviors: Cognitive Dietary Restraint, Disinhibited Eating, and Predisposition to hunger. Cognitive restraint was the domain of highest interest for this study and is reported here. Higher scores in each domain indicate more of each of those behaviors.
  The cognitive restraint domain score is calculated by taking the average of the 21 items in that domain. Each of the 21 items has a score of 0 or 1.
  MINIMUM mean score for this measure is: 0 and MAXIMUM mean score is 1. MINIMUM total score for this measure is: 0 and MAXIMUM total score is 21 (relevant to the "Full Range" in the data table below)
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | -0.83 [-7 to 5] | -0.33 [-7 to 3]

24. Secondary Outcome: Change in Total Weight Related Quality of Life- Adolescent/Young Adult Report
Description: "Impact of Weight on Quality of Life-Kids" questionnaire will be completed by the adolescents age <=19.
  Total and each of the 4 sub scales (Physical Comfort-6 items, Body Esteem-9 items, Social Life-6 items, and Family Relations-6 items) range from a minimum score of 0 to a maximum of 100.
  Higher scores indicate higher quality of life.
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: units on a transformed scale
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
units on a transformed scale | -0.38 [-6.48 to 7.41] | 3.61 [-8.33 to 17]

25. Secondary Outcome: Change in Total Weight Related Quality of Life- Parent Reported of Adolescent/Young Adult
Description: "Impact of Weight on Quality of Life-Kids Parent Proxy" questionnaire will be completed by the parent of the adolescent/young adult.
  Total and each of the 4 sub scales (Physical Comfort-6 items, Body Esteem-9 items, Social Life-6 items, and Family Relations-6 items) range from a minimum score of 0 to a maximum of 100.
  Higher scores indicate higher quality of life.
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: units on a transformed scale
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
units on a transformed scale | 4.94 [0.92 to 12.96] | -0.62 [-15.74 to 25]

26. Secondary Outcome: Change in General Health Related Quality of Life: Total Score PedsQL Instrument - Self Report
Description: PedsQL instrument will be completed by the adolescent/young adult. The CHANGE in total scale score is reported here. The total scale score at each time point ranges from a MIN of 0 to a MAX of 100.
  Items are rated on a 0-4 scale. Items are reverse scored and linearly transformed to a 0-100 scale, such that 0=100, 1=75, 2=50, 3=25, and 4=0.
  Scale Scores are calculated as the sum of the items over the number of items answered.
  Higher scores indicated better health-related quality of life.
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: units on a transformed scale
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
units on a transformed scale | -3.67 [-18 to 7] | 3.17 [-18 to 18]

27. Secondary Outcome: Change in Depression
Description: The adolescent/young adult will complete the 20-item Center for Epidemiologic Studies Depression Scale (CES-D).
  Each item is rated on a 0 to 3 scale (positive items are reverse scored). Minimum score is 0 and maximum is 60. Higher scores indicate more depressive symptoms. Total score is calculated by summing each of the 20 individual items scores.
Time Frame: Baseline and 12 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 6 | 6
units on a scale | 6.5 [1 to 15] | -2.5 [-11 to 5]

28. Secondary Outcome: Participant Satisfaction: Questionnaire
Description: The participating family will be asked to complete a satisfaction questionnaire that will assess reasons for participation, experience during study visits, satisfaction with the effect of the study drug, ease of communication with study staff, and study burden.
  The outcome presented here is the average of the parent and adolescent/young adult dyad's response to the statement: "My overall experience was positive" [1=Strongly disagree, 5=Strongly agree]
Time Frame: At 12 weeks
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Phentermine & Topiramate | Placebo
Number analyzed (Participants) | 12 | 12
units on a scale | 4.75 [4.5 to 5] | 4.75 [4 to 5]

ADVERSE EVENTS:
Time Frame: Adverse event data for the entire trial were collected from the first study activity of the first participant through the final study activity of the last participant, which was from: 2/10/20 through 1/25/22. In general, for each participant, adverse event screening lasted from the enrollment visit through the final study phone call (~4 months).
Arm/Group | Phentermine & Topiramate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phentermine & Topiramate (N=6) | Placebo (N=6)
Hospital admission (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Severe back pain, which after inpatient diagnostic evaluation was deemed not to be related to study intervention. Specifically, no evidence of nephrolithiasis was found.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Phentermine & Topiramate (N=6) | Placebo (N=6)
Restlessness (General disorders) | 6 | 2
Depressed mood (Psychiatric disorders) | 4 | 3 — subjectively reported as different from baseline
Difficulty with sleep (General disorders) | 4 | 3
Fatigue (General disorders) | 5 | 2
Irritability (Psychiatric disorders) | 6 | 1
Paresthesias (Nervous system disorders) | 6 | 1
Anxiety (Psychiatric disorders) | 5 | 1 — subjectively reported - above baseline
Difficulty with concentration/attention (Nervous system disorders) | 5 | 1
Nausea/Vomiting (Gastrointestinal disorders) | 4 | 2
Change in Taste (Gastrointestinal disorders) | 3 | 2
Eye discomfort (Eye disorders) | 1 | 4
Flushing (General disorders) | 4 | 1
Memory problems (Nervous system disorders) | 4 | 1
Menstruation change (Reproductive system and breast disorders) | 2 | 3/4 — Among participants with biological sex of female
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 3
Mental fogginess (Nervous system disorders) | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Word finding difficulties (Nervous system disorders) | 3 | 1
Back, side, and/or groin pain (Musculoskeletal and connective tissue disorders) | 3 | 0
COVID disease (Infections and infestations) | 1 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 2
Fever (Infections and infestations) | 2 | 1
Blurry vision (Eye disorders) | 1 | 1
Decreased sweating (General disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Myalgias (Musculoskeletal and connective tissue disorders) | 0 | 2
Palpitations (Cardiac disorders) | 2 | 0
Esophageal fullness (Gastrointestinal disorders) | 1 | 0
Finger fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Inability to cool down (General disorders) | 1 | 0
Swelling in arms, legs, face (General disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Vaginal pain (Reproductive system and breast disorders) | 1 | 0/4 — Among female participants (mentioned under "any other adverse event experienced")
Depression Score by CES-D that increased from normal to elevated (>=20) on study (Psychiatric disorders) | 3 | 2
Suicidality screen (CSSRS) positivity on study (Psychiatric disorders) | 0 | 0
Low bicarbonate (<20mmol/L) (Metabolism and nutrition disorders) | 3 | 0
Low potassium (<3.5mmol/L) (Metabolism and nutrition disorders) | 1 | 0
Elevated creatinine (Renal and urinary disorders) | 1 | 0 — above upper limit of normal mg/dL
Positive urine pregnancy test (Pregnancy, puerperium and perinatal conditions) | 0 | 0/4 — Among female participants
Elevated systolic blood pressure (>=120mmHg) (Cardiac disorders) | 3 | 2 — at any visit while on study treatment
Elevated diastolic BP (>=80mmHg) (Cardiac disorders) | 1 | 3 — at any visit while on study treatment
Elevated heart rate (>=100 beats per minute) (Cardiac disorders) | 0 | 0 — at any visit while on study treatment
Elevated temperature (measured) (General disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT04095104/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT04095104/ICF_001.pdf